CLINICAL TRIAL: NCT02334254
Title: Rivaroxaban in Patients With Atrial Fibrillation and Coronary Artery Disease Undergoing Percutaneous Coronary Intervention
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yujie Zhou, Vice President of Beijing Anzhen Hospital, Capital Medical University, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: anzhen2013009
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Atrial Fibrillation
Keywords: safety; rivaroxaban; ticagrel; triple antithrombotic regimen; undergoing PCI
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban; Warfarin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dual antithrombotic therapy (DAT) (Experimental): Dual Antithrombotic Therapy (DAT) regimen of rivaroxaban 2.5mg/5mg b.i.d. plus ticagrelor 90mg b.i.d.
  Interventions: Drug: rivaroxaban and ticagrel therapy
- Triple antithrombotic therapy (TAT) (Active Comparator): Triple antithrombotic therapy (TAT) regimen of aspirin 100mg q.d., clopidogrel 75mg q.d. plus warfarin (INR 1.8-2.5).
  Interventions: Drug: triple antithrombotic regimen with warfarin, asipirin and clopidogrel

INTERVENTIONS:
Drug: rivaroxaban and ticagrel therapy — Antiplatelet therapy are mandatory at least 1 month after bare metal stent implantation, and 6 months after drug-eluting stent implantation.
  Arms: Dual antithrombotic therapy (DAT)
Drug: triple antithrombotic regimen with warfarin, asipirin and clopidogrel
  Arms: Triple antithrombotic therapy (TAT)

SUMMARY:
To evaluate the safety for the combination of Rivaroxaban and Ticagrel versus triple antithrombotic regimen (Vitamin K Antagonist (VKA), Clopigogrel and Aspirin) in patients with atrial fibrillation and coronary artery disease undergoing percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
This is an open-label (both physician and participant know the treatment that the participant receives), randomized (study medication is assigned by chance), multicenter clinical study assessing the safety of the combination of rivaroxaban and ticagrel versus triple antithrombotic regimen (warfarin, clopigogrel and aspirin) in patients, who have paroxysmal, persistent, or permanent non-valvular atrial fibrillation (AF) and concomitant coronary artery disease undergoing percutaneous coronary intervention (PCI). A target of 420 participants will be randomized into the study, with approximately 210 participants in each treatment strategy group. Primary comparisons will be made of the rates of major and clinically relevant bleeding, assessed by the modified International Society of Thrombosis and Haemostasis (ISTH) classification. The study consists of a screening phase, a 12-month open-label treatment phase, and an end-of-treatment/early withdrawal visit. The total duration of participation in the study for each participant is approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

* a long-term indication for oral anticoagulation treatment (until at least 1 year after the study)
* a severe coronary lesion (at least 75% stenosis on angiography or fractional flow reserve lower than 0•80) with indication for PCI
* age 18-80 years

Exclusion Criteria:

* history of intracranial bleeding;
* cardiogenic shock;
* contra indication to use of antiplatelet or anticoagulation drugs;
* peptic ulcer in the previous 6 months;
* thrombo cytopenia (platelet concentration lower than 50~10⁹/L);
* major bleeding (according to the Thrombolysis in Myocardial Infarction [TIMI] criteria) in the past 12 months; and
* pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Major or clinically relevant non-major bleeding | 12 months
  Major bleeding was assessed by the International Society of Thrombosis and Hemostasis (ISTH) definition. It included bleeding that was fatal, occurred in a critical location (intracranial, intraspinal, intraocular, retroperitoneal, intraarticular, intramuscular with compartment syndrome, or pericardial), or was associated with a fall in hemoglobin of 2 g/dL or a transfusion of 2 units of packed red blood cells. Clinically relevant non-major bleeding was defined as bleeding that required medical or surgical intervention.

SECONDARY OUTCOMES:
Composite outcome of death, myocardial infarction, stent thrombosis and ischemic stroke | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yujie Zhou, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital,Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Gao F, Shen H, Wang ZJ, Yang SW, Liu XL, Zhou YJ. Rationale and design of the RT-AF study: Combination of rivaroxaban and ticagrelor in patients with atrial fibrillation and coronary artery disease undergoing percutaneous coronary intervention. Contemp Clin Trials. 2015 Jul;43:129-32. doi: 10.1016/j.cct.2015.05.012. Epub 2015 May 21. PMID 26003433